CLINICAL TRIAL: NCT03026660
Title: Effect of Moringa Oleifera on Bone Density in Post-Menopausal Women
Brief Title: Moringa Oleifera on Bone Density
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Appalachian State University (Other)
Collaborators: North Carolina Agriculture & Technical State University (Other)
Responsible Party: Principal Investigator, Edward Merritt, Assistant professor, Appalachian State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 15-0257
Record Dates: First submitted 2017-01-16; First posted 2017-01-20 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Osteoporosis, Osteopenia; Postmenopausal Osteoporosis
Keywords: Moringa Oleifera
MeSH Terms: conditions — Osteoporosis; Bone Diseases, Metabolic; Osteoporosis, Postmenopausal | interventions — flocculant protein MO 2.1, Moringa oleifera

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moringa treatment (Experimental): Moringa Oleifera was distributed in two 500mg capsules of dried and powdered Moringa Oleifera leaves. Two capsules were taken daily.
  Interventions: Dietary Supplement: Moringa Oleifera
- Placebo (Placebo Comparator): The placebo consisted of dried and powdered cabbage in two 500mg capsules. Two capsules were taken daily.
  Interventions: Dietary Supplement: Cabbage Placebo

INTERVENTIONS:
Dietary Supplement: Moringa Oleifera
  Arms: Moringa treatment
Dietary Supplement: Cabbage Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the effects of Moringa Oleifera on the structure and function of bone in post-menopausal women ingesting 1000 mg of Moringa Oleifera daily for 12 weeks.

DETAILED DESCRIPTION:
Moringa Oleifera (M. Oleifera) is a tropical plant native to northern India, Pakistan, Himalayan regions, Africa, Central America, and Arabia that has been used for centuries in ethnic cultures all over the world. M. Oleifera is exceptionally rich in a variety of nutrients and medicinal phytochemicals, including those that promote bone density, such as vitamin D, calcium, phosphorus, magnesium and others. M. Oleifera also contains micronutrients that play a critical role in bone health and in calcium absorption, such as boron, vitamin C, magnesium, potassium, phosphorous and others. For instance, boron stabilizes and extends the half-life of vitamin D; magnesium (Mg) affects the activities of osteoblasts and osteoclasts, as well as bone homeostasis by modulating the concentration of parathormone and the activated form of vitamin D. Magnesium also contributes to bone structural development; vitamin K reduces bone turn over, improves bone strength and plays an essential role in osteocalcin carboxylation and vitamin C increases bone density and strength by increasing collagen formation and promotes healing during fracture. Collectively, these micronutrients in M. Oleifera are expected to significantly impact bone health. Given this knowledge, the purpose of the present study is to determine the effects of M. Oleifera on the structure and function of bone in post-menopausal women ingesting 1 gram of M. Oleifera daily for 12 weeks using DEXA scans.

The fresh young leaves of Moringa oleifera (about 2 years old) were collected by Dr. Joshua Idassi, from a field and high tunnel plots at the North Carolina Agriculture and Technical State University farm in July, 2014. Botanical identification and authentication were performed by Dr. Joshua Idassi, Natural Resources Specialist, from the Cooperative Extension Program, North Carolina A & T. A voucher specimen (LUH 2923) was deposited in the herbarium of the University of Lagos, Akoka, Yaba, Lagos. Fresh leaves of M. Oleifera were air-dried for about 7 days at 30 ◦C and macerated into a fine powder.

Twenty-four untrained post-menopausal women (60-70 years old) were randomly assigned to either the control or placebo group (no program) or the experimental /treatment group (M. Oleifera supplement group). Both groups orally ingested 1 gram (1000 mg) daily of cabbage (placebo) or M. Oleifera (treatment group) leaf powder in capsules for 12 weeks. The bone scans were then taken pre-supplementation and after 12 weeks to determine the effects of M. Oleifera on various bone parameters, including bone mass density, bone mineral content, and select anthropomorphic results including weight, body fat percentage, and lean mass percentage.

The first visit to the laboratory by participants was utilized for providing them with general information and as a testing session. Specifically, the information session consisted of educating them on and obtaining signatures for informed consent, and conducting health history and physical activity questionnaire. The first testing session consisted of obtaining the pre-supplementation DEXA scans. The participants were then given six weeks' worth of their supplement. The subjects came back to the testing site again at six weeks (midway of supplementation) to pick up their supplement for the last six weeks and were then instructed on how to fill out a three-day diet log. The diet log was analyzed and averaged using the USDA Super Tracker online program. The third and last visit was 12 weeks after the start of supplementation and during this visit the second set of DEXA scans were obtained and the diet records were obtained. These records were used to determine the normal diet nutrients as well as caffeine intake of the participants.

DEXA scanning allows for the measurement of whole body bone density, as well as the specific density of the hip and femoral head. The subjects were laid on the DEXA machine scanner motionless for 6-10 minutes while the scan was performed. The first scan measured total body bone density, as well as the basic body composition. The subject were then asked to lay motionless for another 6-10 minutes while another DEXA scan was completed, which measured the bone density and characteristics of the hip and femoral head.The BMD, t-score and z-scores of the whole body were recorded, as well as the BMD, t-score, and z-scores of the right and left total hip and femoral necks. These data points were used to determine whether there were any significant differences between the two groups after the intervention period.

The supplementation of the M. Oleifera was began after the first visit which included the signing of the consent form, the performance of the pQCT and the DEXA scans. Once the subjects were scanned they (subjects) were randomly assigned to either the placebo or the M. Oleifera group. The M. Oleifera group was given the whole leaf M. Oleifera powder in capsule form at 1000mg daily for 12 weeks and similarly the control group was given the same amount of cabbage powder in capsule form and route. However, the placebo capsule consisting of cabbage had significantly lower levels of vitamins and nutrients compared to M. Oleifera. M. Oleifera was harvested and processed under optimal conditions and was carefully weighed on a scale and packed into capsules under sterile conditions. Each capsule for both groups contained 500 mg of the supplement, implying that each participant regardless of their weight took two capsules daily orally for 12 weeks. If they missed a day they were instructed not to double the dosage the next day. The placebo group was given the exact same instructions for consumption as the M. Oleifera group, and the study was conducted in a double blind manner. The dietary records were collected and analyzed to determine any significant differences between the two groups based on normal daily consumed nutrients.

ELIGIBILITY:
Inclusion Criteria:

* Between 60 -70 years old
* Female

Exclusion Criteria:

* Fracture in non-dominant forearm/wrist or lower leg.
* Currently taking blood thinners
* Currently taking estrogen supplements
* Have had a hysterectomy

Ages: 60 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Females only
Enrollment: 20 (Actual)
Dates: Start 2015-07; Primary Completion 2016-02 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Bone Density | 12 weeks after start of intervention
  Measured by Dual Energy X-Ray Absorptiometry

CONTACTS AND LOCATIONS:
Overall Officials: Edward K Merritt, PhD, Principal Investigator — Appalachian State University
Locations (1):
- Appalachian State University, Boone, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burge R, Dawson-Hughes B, Solomon DH, Wong JB, King A, Tosteson A. Incidence and economic burden of osteoporosis-related fractures in the United States, 2005-2025. J Bone Miner Res. 2007 Mar;22(3):465-75. doi: 10.1359/jbmr.061113. PMID 17144789
- [Background] Popoola JO, Obembe OO. Local knowledge, use pattern and geographical distribution of Moringa oleifera Lam. (Moringaceae) in Nigeria. J Ethnopharmacol. 2013 Nov 25;150(2):682-91. doi: 10.1016/j.jep.2013.09.043. Epub 2013 Oct 2. PMID 24096203
- [Background] Thurber MD, Fahey JW. Adoption of Moringa oleifera to combat under-nutrition viewed through the lens of the "Diffusion of innovations" theory. Ecol Food Nutr. 2009 May-Jun;48(3):212-25. doi: 10.1080/03670240902794598. PMID 20161339
- [Background] Singh V, Singh N, Pal US, Dhasmana S, Mohammad S, Singh N. Clinical evaluation of cissus quadrangularis and moringa oleifera and osteoseal as osteogenic agents in mandibular fracture. Natl J Maxillofac Surg. 2011 Jul;2(2):132-6. doi: 10.4103/0975-5950.94466. PMID 22639499
- [Background] Zeng FF, Xue WQ, Cao WT, Wu BH, Xie HL, Fan F, Zhu HL, Chen YM. Diet-quality scores and risk of hip fractures in elderly urban Chinese in Guangdong, China: a case-control study. Osteoporos Int. 2014 Aug;25(8):2131-41. doi: 10.1007/s00198-014-2741-2. Epub 2014 May 27. PMID 24861906
- [Background] Storm D, Eslin R, Porter ES, Musgrave K, Vereault D, Patton C, Kessenich C, Mohan S, Chen T, Holick MF, Rosen CJ. Calcium supplementation prevents seasonal bone loss and changes in biochemical markers of bone turnover in elderly New England women: a randomized placebo-controlled trial. J Clin Endocrinol Metab. 1998 Nov;83(11):3817-25. doi: 10.1210/jcem.83.11.5289. PMID 9814452
- [Background] Nandave M, Ojha SK, Joshi S, Kumari S, Arya DS. Moringa oleifera leaf extract prevents isoproterenol-induced myocardial damage in rats: evidence for an antioxidant, antiperoxidative, and cardioprotective intervention. J Med Food. 2009 Feb;12(1):47-55. doi: 10.1089/jmf.2007.0563. PMID 19298195